CLINICAL TRIAL: NCT02569736
Title: Characterization of the Effect of Tocilizumab in Vivo and in Vitro on T Follicular Helper Cells in Rheumatoid Arthritis Patients and Consequence on B Cells Maturation
Acronym: Tocihelper
Status: Completed | Type: Observational
Sponsor: Association Aquitaine de Recherche Clinique en Rhumatologie (Other)
Collaborators: Roche Pharma AG (Industry); Chugai Pharma France (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29237
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Arthritis, Rheumatoid; Tocilizumab; T-Lymphocytes, Helper-Inducer
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tocilizumab: Patients with active moderate to severe RA fulfilling ACR criteria and requiring TCZ treatment, according to the EU label and French authority recommendations, who accept to enter the study and to sign the informed consent.
- Methotrexate: Patients with active moderate to severe RA fulfilling ACR criteria and requiring MTX treatment, according to the EU label and French authority recommendations, who accept to enter the study and to sign the informed consent.
- Healthy Controls: Healthy controls will be defined as people non-affected by an inflammatory disease (such as RA, ankylosing spondylitis, lupus…). This group will be constituted with patients affected by sciatica, osteoarthritis, osteoporosis…

SUMMARY:
Naïve CD4+ helper T (Th) cells, upon encountering their cognate antigens presented on professional antigen-presenting cells, differentiate into different effector cells:

* Th1 cells produce Interferon-γ and regulate antigen presentation and immunity against intracellular pathogens;
* Th2 cells produce IL-4 (Interleukin-4), IL-5 and IL-13, and mediate humoral responses and immunity against parasites;
* Th17 cells produce IL-17, IL-17F and IL-22 and regulate inflammatory responses by tissue cells.

An additional TH subset called follicular helper T (Tfh) cells has recently been identified in germinal centers and also in whole blood (circulating Tfh cells). These cells regulate B-cell maturation and immunoglobulin production during normal immune responses. They produce factors essential for B cell selection and maturation into memory B-cells or long-lived antibody-secreting plasma cells. Furthermore, they also seem to favor pathogenic autoantibody production in systemic autoimmunity, and therefore could potentially represent a novel therapeutic target in autoimmune diseases. Indeed, rheumatoid arthritis synovium is characterized by the presence of ectopic lymphoid structures, resembling germinal centers. Potentially, Tfh cells from these nonlymphoid tissues could promote B-cell maturation and synthesis of pathogenic autoantibody production, thus potentiating tissue injury. Interestingly, production of IL-21 by Tfh cells is implicated in B cell activation, and the same cytokine have been associated with rheumatoid arthritis (RA) pathogenesis.

IL-6 blocking therapy significantly reduces signs and symptoms as well as radiological progression in RA. However, so far, it has not been determined which of the pleiotropic IL-6 effects impact the observed clinical response. Recently, Samson et al have demonstrated that Tocilizumab (TCZ) corrects the imbalance between Th17 cells and Treg cells in patients with RA. More interestingly, the group of Hans-Peter Tony has reported the impact of TCZ on B cell compartment. They showed a significant reduction in the frequency of peripheral pre-switch and post-switch memory B cells but also a reduction of serum immunoglobulin levels, that could be the reflect of TCZ on Tfh cells development, circulation and/or function.

Most of the work studying the role of IL-6 on Tfh cells development has been performed in mice. They showed that optimal Tfh cells formation requires IL-21 and IL-6, and that cytokines alone are insufficient to drive Tfh cells differentiation.

To better understand the impact of IL-6 on human Tfh cells, the investigators would like to conduct a prospective study in patients with active RA and investigated the effects of blocking IL-6 with TCZ on circulating Tfh cells levels and Tfh cells subsets over a 12-week study period. Furthermore, the impact of TCZ treatment on Tfh cells generation will be explored in vitro.

ELIGIBILITY:
Inclusion Criteria:

Inclusion in TCZ and MTX groups:

* Patients with active moderate to severe RA fulfilling ACR criteria and requiring TCZ or MTX treatment, according to the EU label and French authority recommendations, who accept to enter the study and to sign the informed consent.
* Patients > 18 years
* When treated with corticosteroids: Dose ≤10mg/jour within 4 weeks before inclusion and dose stable during the study.
* When treated with MTX (0.3 mg/kg/w): Dose stable within 4 weeks before inclusion and during the study to avoid confusion on Tfh levels evaluation.
* When treated by prior anti-TNF: according to the recommendations of the French "Club Rhumatismes Inflammatoires", a wash-out period of 5 half-lives will be defined to avoid confusion in the evaluation of Tfh cells initial levels.
* These patients will be consecutively included in the study until the number of needed patients will be reached.

Inclusion in the healthy controls group:

* Healthy controls will be defined as people non-affected by an inflammatory disease (such as RA, ankylosing spondylitis, lupus…). This group will be constituted with patients affected by sciatica, osteoarthritis, osteoporosis…
* These patients will be included in a second phase in order to guarantee the quality of matching with cases.

Exclusion Criteria:

* Patients previously treated with TCZ
* Patients with a history of allergic reactions or Hypersensitivity to TCZor to any of the excipients
* Patients with severe and uncontrolled infections such as sepsis and opportunistic infections
* Patients with hepatitis B (with virus replication) or C, HIV-infection and tuberculosis
* Patients with history of cancer or lymphoma
* Patients with history of diabetes
* Patients who presented one of the following laboratory abnormalities:

  * Serum creatinine > 1.6 mg/dL (141 μmol/L) in female patients and > 1.9 mg/dL (168 μmol/L) in male patients, only for MTX treated patients.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN).
  * Platelet count < 100,000/mm3, (100 x 109/L).
  * Hemoglobin < 8.0 g/dL, (5.0 mmol/L).
  * White Blood Cells < 3000/mm3, (3.0 x 109/L).
  * Absolute neutrophil count < 2000/mm3, (2.0 x 109/L).
  * Absolute lymphocyte Count < 500/mm3, (0.5 x 109/L).
  * Positive hepatitis BsAg or hepatitis C antibody
  * Total bilirubin > ULN
* Pregnant or breast-feeding patients
* Patients who refuse to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be performed as a prospective observational open-labeled study (non-interventional) to evaluate the impact of TCZ treatment on the evolution of circulating Tfh cells levels. The administration of treatments (TCZ and MTX) will be done according to current practice, and will not be motivated by the inclusion in this study. TCZ will be administered in association with a conventional DMARD, or in monotherapy, according to clinical recommendations. The objective of this study is to analyze the impact of new therapy set-up, and patients included in the TCZ group would be under MTX treatment for at least 3 months. The immunological analysis will be performed with drop-off of blood samples used in the recommended follow-up of patients treated by MTX or TCZ. For the healthy controls, the immunological analysis will be performed with drop-off of blood samples used in the recommended follow-up of patients treated for osteoporosis or osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in levels of circulating Tfh cells at 12 weeks for TCZ treated patients | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology department - Bordeaux University Hospital, Bordeaux, Aquitaine, France